CLINICAL TRIAL: NCT00360256
Title: Pharmacogenetic Study of CYP450 2D6 and 2C19 in Patients With Significant Adverse Effects From Antidepressants
Brief Title: Genetic Study of Liver Enzymes in Patients With Side Effects From Antidepressants
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Zixuan Wang, Ph.D., Medical College of Georgia
Other Study IDs: CYP450 Antidepressant study; HAC File #: 06-04-278
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Amplichip P450 tests; Antidepressants
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control
- Case group

SUMMARY:
The objective of this pilot study is to determine the genetic polymorphism rate of CYP450 2D6 and 2C19 metabolic enzymes in patients with significant adverse effects from antidepressants, compared to a population of patients who had no significant adverse effects from antidepressants metabolized by CYP2D6 and 2C19.

The hypothesis for the proposed research is that the rate of 2D6 and 2C19 alleles that are associated with poor metabolizer status in the treatment-intolerant population will far exceed the rate found in patient population who takes antidepressants without adverse effects.

DETAILED DESCRIPTION:
Study Design This is a naturalistic study of sixty patients, which will include 30 patients who had side significant adverse reactions from treatment with antidepressants metabolized by CYP2D6 and 2C19 (TREATMENT-INTOLERANT group) and 30 patients who responded to treatment with same group of antidepressants without significant adverse effects (CONTROL group). The study is expected to last for one year.

Once recruitment, subject consent, and competency to participate have been achieved, the diagnosis will be assessed through clinical interview, aided by medical records, when available. A complete medication history will be taken including all known medications, their doses, and duration of use, to determine exposure to antidepressants metabolized by CYP450 2D6 and 2C19 and absence of concomitant CYP 2D6 and 2C19 inhibitors. A list of the antidepressants metabolized by CYP450 2D6 and 2C19 and their inhibitors is attached. If exposure is confirmed, each subject will be interviewed using the English version of UKU (Udvalg for Kliniske Undersogelser) Rating Scale14 to retrospectively assess their side effects from medications metabolized by CYP 2D6 and 2C19 enzymes. We will use the modules 1, 3 and 4 of the UKU, for "psychic", "autonomic" and respectively "other" side effects. Only patients who had marked side effects from one medication or either moderate or marked side effects from two medications metabolized by CYP 2D6 and 2C19 enzymes, according with UKU, will be included in the TREATMENT-INTOLERANT group. Subjects who have none or mild adverse effects, will be included in the CONTROL group. The subject interview is expected to last approximately ninety minutes and will be conducted by a sub investigator (Adriana Foster, MD).

The study participants will be asked to rinse mouth with water to remove food particles and spit saliva into a collection cup until the liquid level reaches the line indicated on the container (~2ml). We will use Oragene ™ DNA self-collection kit (DNA Genotek, Inc, Ottawa, Ontario, Canada).

The saliva will be transported to GEM Labs, located on MCG campus, by research staff. The genomic DNA will be extracted with the reagent and method supplied by the manufacturer, Oragene. This will be used as the template to amplify the relevant regions of CYP450 2D6 and 2C19. The PCR products will be randomly cleaved into 50 to 100 bp by digestion with DNase I. These fragments will be further labeled with phycoerythrin (PE), a fluorescent dye. The PE labeled fragments will be hybridized to the P450 Roche AmpliChip, washed, and scanned by the Affymetrix automated GeneChip fluidics Station 450Dx and the Affymetrix GeneChip scanner 3000Dx with GeneChip Operating Software Dx 1.1.3. The data will be analyzed by AmpliChip CYP450_US Data Analysis to determine the genotype for 2D6 (it totally assesses 27 mutation sites, deletion, and duplication) and 2C19 (2 mutation sites). Genotyping results will be analyzed by the same software to predict the phenotype (ultra rapid, extensive, intermediate, and poor metabolizer).

Overall, the study requires only one visit from the participant; after interviewing and saliva sample have been completed, the participant's role in the research will be fulfilled. This study will be carried out in its entirety at the Medical College of Georgia facilities. We hope to demonstrate that the rate of 2D6 and 2C19 alleles that are associated with poor metabolizer status in the treatment-intolerant population will far exceed the rate found in patient population who takes antidepressants without adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between ages 18 and 65 of any ethnic background
* Diagnosis of major depressive disorder, dysthymic disorder or depressive disorder NOS.
* Experienced side effects on antidepressant metabolized by CYP 2D6 and 2C19 that required discontinuation of treatment
* Experienced side effects from 2 or more antidepressants metabolized by CYP 2D6 and 2C19

Exclusion Criteria:

Exclusion criteria:

* Patients with diagnosis of bipolar disorder or any anxiety disorder. We decided to exclude patients with these diagnoses, due to the fact that antidepressants may exacerbate symptoms of bipolar and anxiety disorders and there is a risk that these symptoms can be attributed instead to antidepressant adverse effects.
* Patients taking inhibitors of drugs metabolized by CYP 2D6 and 2C19
* Patients who are non-English speaking: the English version of the UKU side effects rating scale will be used. The rating of side effects depends on the patient interview and the information found in the medical record. To appreciate the extent of the side effects, the rater and the research participant must be speaking the same language. Thus, to include non-English speaking participants, both the research and the clinical staff would need to be fluently bilingual, which is not the case at MCG inpatient and outpatient treatment facilities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Depressed patients
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Cytochrome P450 2D6 and 2C19 genotype | 12/07

SECONDARY OUTCOMES:
Drug tolerability | December 2007

CONTACTS AND LOCATIONS:
Overall Officials: Adriana E. Foster, M.D., Study Director — Assistant Professor of Psychiatry MCG; Zixuan Wang, Ph.D., Principal Investigator — Assistant Research Scientist MCG Dept of Pathology
Locations (1):
- Medical College of Georgia, Dept. of Psychiatry and Health Behavior, Augusta, Georgia, United States